CLINICAL TRIAL: NCT05382078
Title: Effectiveness and Safety Evaluation of Nafamostat Mesilate During Continuous Renal Replacement Therapy in Critically Ill Patients
Brief Title: Nafamostat Mesilate for Anticoagulation During CRRT in Critically Ill Patients
Acronym: NMFADCICIP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Second Affiliated Hospital of Xi'an Jiaotong University (Other); Tang-Du Hospital (Other); Xi'an Gaoxin Hospital (Other); Affiliated Chest Hospital Xi'an Jiaotong University (Unknown); Xi'an Honghui Hospital (Other); Shangluo Central Hospital (Other); Yulin first Hospital (Unknown); Yan'an University Affiliated Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2022LSK-202
Record Dates: First submitted 2022-05-07; First posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-04

CONDITIONS: Sepsis Syndrome; MODS; AKI; Hemorrhage; Trauma; Thrombus
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome; Multiple Organ Failure; Hemorrhage; Wounds and Injuries; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Continuous renal replacement therapy is widely used in intensive care medicine, which is known as an alternative therapy to save injured kidney . Anticoagulation is an important part of this therapy. An insufficient anticoagulation would cause a poor curative effect of CRRT. Hemorrhage，heparin-induced thrombocytopenia (HIT), citrate accumulation, acidosis ad filter extra-cost usually happened on anticoagulation during CRRT. Therefore a new effective anticoagulation of CRRT needs to be carried out. Nafamostat Mesylate (NM) is a new anticoagulant. This serine protease inhibitor with broad spectrum can inhibit kinds of enzymes on the process of coagulation. NM is mainly rapidly decomposed in the liver and also removed by dialysis or filtration. The elimination half life of is only 8 minutes. If NM is applied as a regional anticoagulant, approximate 40% NM is removed by dialysis and / or convection in cardiopulmonary bypass circuit, and then rapidly degraded by esterase in liver and blood, which ensures security in patients with bleeding tendency.

Based on the information above, the investigators designed an observational clinical study aimed to testify that NM would have equivalent anticoagulant results compared with those traditional ways and might even have a better effect than traditional anticoagulant therapy.The study team has investigated the current situation of CRRT in Shaanxi province in China through a cross-sectional survey last year. The survey involved 74 hospitals in Shaanxi province and the results basically illustrated a real status of CRRT. These scientific results helped investigators to design this multi-center, parallel, controlled, non intervention study and real world study.

DETAILED DESCRIPTION:
CRRT, the continuous renal replacement therapy, is widely applied in the field of intensive care medicine. This technology is known as an alternative therapy to save injured kidney with advantages of the accurate volume control, stable acid-alkali electrolyte equilibrium maintenance and hemodynamic stability.

Anticoagulation is an important part of this therapy. An ideal anticoagulant and a reasonable anticoagulation process would help CRRT function well. Therefor an insufficient anticoagulation would cause a poor curative effect of CRRT.

Heparins, reginal citrate anticoagulant (RCA) and anticoagulant-free are the most common methods applied in CRRT. However, heparins would lead to hemorrhage and heparin-induced thrombocytopenia (HIT). And RCA is the absolute contraindication of liver failure and shock status, which would easily cause citrate accumulation and acidosis. While anticoagulant-free method is often suitable for patients with acute hepatic failure, citrate metabolic disorder, sever acidosis and coagulation dysfunction. According to aforementioned reasons, a new effective anticoagulation of CRRT needs to be carried out.

Nafamostat Mesylate (NM) is a late-model anticoagulant. This serine protease inhibitor with broad spectrum can inhibit kinds of enzymes on the process of coagulation. It has strong inhibitory effects on thrombin, coagulation factors Ⅻ a, Xa, VIIa, kallikrein, fibrinolytic enzyme, complement system C1r, C1s and trypsin. NM is mainly rapidly decomposed by carboxylesterase in the liver and also removed by dialysis or filtration. The elimination half life of is only 8 minutes. If NM is applied as a reginal anticoagulant, approximate 40% NM is removed by dialysis and / or convection in cardiopulmonary bypass circuit, and then rapidly degraded by esterase in liver and blood, which ensures security in patients with bleeding tendency.

Based on the information above, the investigators designed an observational clinical study aimed to testify that NM would have equivalent anticoagulant results compared with those traditional ways and might even have a better effect than traditional anticoagulant therapy.

In this study, the average filter life-span will be calculated and compared in groups to assess effectiveness of NM. And the safety of NM will be assessed by comparing the incidence rate of the bleeding and/or massive hemorrhage between groups. Besides, the best dose of NM will be titrated during the trial along with targeting a best monitoring value of NM.

Either in the observational or in the control group, the continuous renal replacement therapy should be implemented as indications. The investigators need to record trial details into an eCRF as protocol required. The details include main diagnosis, clinical status before first CRRT, the primary indications for first CRRT, the coagulation function, laboratory indexes, the frequency and site of hemorrhage, the incidence of hyper-coagulable state, the average life-span of filters during first CRRT, the number of filters caused by clotting, and times of transfusion.

The anticoagulation in observational arm will be implemented as follows.

1. Admixture: to fully dissolve 50mg NM into 5% glucose solution.
2. Pipeline pre-flushing: to dissolve 50mg NM into 1000ml 5% glucose solution. to prime the filters and extracorporeal circuits with the mixtures above. Then to use 5% glucose solution and 0.9% saline solution sequentially flushing the pipe-line and filters for a complete elution and to ensure the drug residue would be as less as possible.
3. Drug infusion: The maintaining dose of NM is 10-20mg/hr.
4. Monitoring: APTT will be tested every 30min to 2h initially. The goal of APTT is settled as 80s-100s in circuits and as 40s-50s in body. Once the steady state is reached, the monitoring interval will be adjusted to 12~24h. To reach the target monitoring goal, the NM will be added or reduced by 2~4mg each time.

While in control group, the CRRT steps will be implemented by Standard operating procedures for blood purification(version2021, China).

Data collection and safety: in this study, an independent offline eCRF will be applied in collecting data. Specific staff will be trained to use eCRF correctly and collect data regularly. The details are displayed in CRF.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patients admitted to ICU
* ICU patients requiring further CRRT due to renal or non-renal indications
* signed informed consent

Exclusion Criteria:

* The hospitalization stay of ICU is less than 24 hours.
* The case data are incomplete.
* age<18 and ≥85
* patients suffering from metal illness or unable to cooperate for some certain reasons
* allergic to NM or Pharmaceutical excipient or extracorporeal circuit consumables
* preparing for pregnancy/pregnant/ during lactation period
* patients or their agents refuse to sign the informed consent form or participate in another clinical trial
* non-compliant, lost visit or other situations that patients are unsuitable for selection determined by researchers

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study plan to enroll 188 cases in 16 intensive care unit in Shaanxi province from January 2022 to December 2024.Patients will be divided into two group based on the anticoagulation method.1)Observation group: using NM as anticoagulant during CRRT；2)Control group: using heparins or RCA or anticoagulant-free during CRRT.
Sampling Method: Probability Sample
Enrollment: 188 (Estimated)
Dates: Start 2022-05-31 (Estimated); Primary Completion 2023-05-04 (Estimated); Study Completion 2024-05-03 (Estimated)

PRIMARY OUTCOMES:
the average filter life-span | up to 96 hours
  The average filter life-span is calculated as the total life-span of filters devided by filter numbers during the first 96 hours of first CRRT. The metric is described as hour per number.

SECONDARY OUTCOMES:
the incidence of bleeding or massive hemorrhage events | From date of first CRRT start until the date of discharge or death, assessed up to 90 days
  This indication is to describe the safety of NM. The incident rate of bleeding or hemorrhage will be counted and calculated to compare the difference between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Qindong Shi, Chief, Study Chair — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xian JiaotongUniversity, Xi'an, Shaanxi, China